CLINICAL TRIAL: NCT00085228
Title: Randomized Phase II Trial of Docetaxel (Taxotere) and Oblimersen (Antisense Oligonucleotide Directed to BCL-2) Versus Taxotere Alone in Patients With Hormone-Refractory Prostate Cancer
Brief Title: Docetaxel With or Without Oblimersen in Treating Patients With Hormone-Refractory Adenocarcinoma (Cancer) of the Prostate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-30021; EORTC-30021; AVENTIS-AVE3139E/2501
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — oblimersen; Docetaxel

INTERVENTIONS:
Biological: oblimersen sodium
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Oblimersen may increase the effectiveness of docetaxel by making tumor cells more sensitive to the drug.

PURPOSE: This randomized phase II trial is studying how well giving docetaxel together with oblimersen works compared to docetaxel alone in treating patients with hormone-refractory adenocarcinoma (cancer) of the prostate.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the activity of docetaxel with or without oblimersen, in terms of prostate-specific antigen response, in patients with hormone-refractory adenocarcinoma of the prostate.
* Compare the toxicity of these regimens in these patients.

Secondary

* Compare the time to progression in patients treated with these regimens.
* Compare survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, metastatic disease (M0 vs M1 with non-measurable lesions only vs M1 with measurable lesions), prior estramustine (yes vs no), and prior bisphosphonates (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive docetaxel IV over 1 hour on day 5 and oblimersen IV continuously on days 1-7.
* Arm II: Patients receive docetaxel IV over 1 hour on day 1. In both arms, treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 8 weeks until progressive disease and then every 16 weeks thereafter.

PROJECTED ACCRUAL: A total of 102 patients (51 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate
* Hormone-refractory disease

  * Disease progression after prior hormonal therapy with luteinizing hormone-releasing hormone (LH-RH) analogues or orchiectomy and antiandrogens (given together or consecutively)
* Prostate-specific antigen (PSA) progression documented by at least 2 increases in PSA values over previous PSA reference value

  * Must demonstrate continued PSA elevation for at least 6 weeks after discontinuation of antiandrogen therapy
* PSA ≥ 5 ng/mL (Hybritech or equivalent) within the past week
* Testosterone ≤ 0.5 ng/mL* NOTE: *Patients with medical castration with LH-RH analogue must continue with LH-RH analogue throughout the study
* No evidence of painful and/or destructive bone metastases requiring concurrent radiotherapy, bisphosphonates, or bone-seeking radionuclides

  * Other bone metastases allowed
* No clinical evidence of brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* WBC ≥ 3,500/mm^3
* Hemoglobin ≥ 10 g/dL

Hepatic

* AST and ALT ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ ULN
* PTT and PT ≤ 1.5 times ULN OR
* INR ≤ 1.3

Renal

* Creatinine ≤ 1.5 times ULN OR
* Creatinine clearance ≥ 50 mL/min

Cardiovascular

* No unstable angina
* No uncontrolled hypertension
* No deep venous thrombosis within the past 6 months
* No cerebrovascular accident, transient ischemic attack, or myocardial infarction within the past 6 months

Pulmonary

* No pulmonary embolism
* No history of interstitial pneumonitis
* No history of pulmonary fibrosis

Other

* Adequate venous access
* HIV negative
* No active infection
* No pre-existing neuropathy
* No hypersensitivity to phosphorothioates
* No hypersensitivity to oligonucleotides or any other component of the oblimersen formulation or to drugs formulated with polysorbate
* No psychological, familial, sociological, or geographical condition that would preclude study compliance
* No other malignancy within the past 5 years except adequately treated superficial urothelial or skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Prior estramustine allowed
* No other prior chemotherapy
* No concurrent estramustine

Endocrine therapy

* See Disease Characteristics
* At least 6 weeks since prior flutamide, bicalutamide, or nilutamide
* More than 6 weeks since prior hormonal manipulation with PC-SPES
* Concurrent LH-RH agonist allowed
* No concurrent antiandrogens

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy involving > 25% of marrow-producing area
* No prior bone-seeking radionuclides
* No concurrent radiotherapy (including palliative therapy for painful bone metastases)
* No concurrent bone-seeking radionuclides

Surgery

* See Disease Characteristics

Other

* Prior bisphosphonates allowed
* No concurrent anticoagulation except for low-dose warfarin (1 mg/day)
* No concurrent regular (daily) intake of opioid analgesics
* No other concurrent experimental drugs or anticancer drugs
* No concurrent bisphosphonates

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2004-04; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Prostate-specific antigen response as measured by Bubley criteria every course until progression or after 12 courses
Severe toxic events as measured by CTCAE v3.0 every course until progression or after 12 courses

SECONDARY OUTCOMES:
Time to progression as measured by RECIST and Bubley criteria every 3 courses, and then every 8 weeks until progression, and every 16 weeks from progression until death
Toxicity as measured by CTCAE v3.0 every 3 courses, and then every 8 weeks until progression, and every 16 weeks from progression until death
Objective response as measured by RECIST every 3 courses, and then every 8 weeks until progression, and every 16 weeks from progression until death
Overall survival as measured by Logrank every 3 courses, and then every 8 weeks until progression, and every 16 weeks from progression until death

CONTACTS AND LOCATIONS:
Overall Officials: Cora N. Sternberg, MD, FACP, Study Chair — Azienda Ospedaliera S. Camillo-Forlanini
Locations (16):
- Kaiser Franz Josef Hospital, Vienna, Austria
- Belgium (5):
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - U.Z. Gasthuisberg, Leuven
- Rigshospitalet - Copenhagen University Hospital, Copenhagen, Denmark
- CHU de Grenoble - Hopital de la Tronche, Grenoble, France
- Assaf Harofeh Medical Center, Ẕerifin, Israel
- Ospedale S. Camillo-Forlanini, Rome, Italy
- Academisch Medisch Centrum at University of Amsterdam, Amsterdam, Netherlands
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- Hospital Desterro, Lisbon, Portugal
- Hospital General Universitari Vall d'Hebron, Barcelona, Spain
- United Kingdom (2):
  - Saint Bartholomew's Hospital, London, England
  - Western Infirmary, Glasgow, Scotland

REFERENCES:
- [Result] Sternberg CN, Dumez H, Van Poppel H, Skoneczna I, Sella A, Daugaard G, Gil T, Graham J, Carpentier P, Calabro F, Collette L, Lacombe D; EORTC Genitourinary Tract Cancer Group. Docetaxel plus oblimersen sodium (Bcl-2 antisense oligonucleotide): an EORTC multicenter, randomized phase II study in patients with castration-resistant prostate cancer. Ann Oncol. 2009 Jul;20(7):1264-9. doi: 10.1093/annonc/mdn784. Epub 2009 Mar 17. PMID 19297314
- [Result] Sternberg CN, Dumez H, Van Poppel H, et al.: Multicenter randomized EORTC trial 30021 of docetaxel + oblimersen and docetaxel in patients (pts) with hormone refractory prostate cancer (HRPC). [Abstract] American Society of Clinical Oncology 2007 Prostate Cancer Symposium, 22-24 February 2007, Orlando, FL. A-144, 2007.